CLINICAL TRIAL: NCT03637374
Title: A Study of the Safety, Efficacy, Longitudinal Costs and Patient-Centered Outcomes Using a TAAA Debranching Device
Brief Title: Safety, Efficacy, Longitudinal Costs and Patient-Centered Outcomes Using a TAAA Debranching Device
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigational device is no longer manufactured
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00075706
Record Dates: First submitted 2018-08-10; First posted 2018-08-20 (Actual); Results first posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-07

CONDITIONS: Thoracoabdominal Aortic Aneurysm
Keywords: aortic aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal; Aortic Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Primary Study Arm (Experimental): The TAAA Debranching Stent Graft System is comprised of two investigational devices including the Visceral Manifold and Thoracic Bifurcation and the unitary manifold. The thoracic bifurcation and the visceral manifold as well as the unitary manifold work to facilitate endovascular stenting of the visceral vessels (renals, celiac, SMA) while maintaining flow to the visceral and infrarenal segments.
  Interventions: Device: Visceral Manifold and Thoracic Bifurcation; Device: Unitary Manifold; Device: TAAA Debranching Stent Graft System
- Expanded Selection Arm (Other): The Expanded Selection Arm will be treated the same as those in the Primary Study Arm. Your doctor will determine what arm you are in. TAAA Debranching Stent Graft System is comprised of two investigational devices including the Visceral Manifold and Thoracic Bifurcation and the unitary manifold. The thoracic bifurcation and the visceral manifold as well as the unitary manifold work to facilitate endovascular stenting of the visceral vessels (renals, celiac, SMA) while maintaining flow to the visceral and infrarenal segments.
  Interventions: Device: Visceral Manifold and Thoracic Bifurcation; Device: Unitary Manifold; Device: TAAA Debranching Stent Graft System

INTERVENTIONS:
Device: Visceral Manifold and Thoracic Bifurcation — Endovascular stent graft system
Device: Unitary Manifold — Endovascular stent graft system
Device: TAAA Debranching Stent Graft System — Endovascular stent graft system

SUMMARY:
The primary purpose of this study is to assess the use of the TAAA Debranching Stent Graft System to repair thoracoabdominal aortic aneurysms in patients having appropriate anatomy, as measured by device safety, effectiveness, costs of delivery of aortic surgery care, and patient quality of life domains. Additionally, the study will assess technical success and treatment success at each follow-up interval.

DETAILED DESCRIPTION:
The primary objective of this clinical investigation is to assess the use of the TAAA Debranching Stent Graft System to repair thoracoabdominal aortic aneurysms. While surgery remains a standard treatment for complex abdominal and thoracoabdominal aneurysms (TAAA), the tolerance of some patients to recover from such extensive and invasive open aortic reconstructions is poor. Endovascular repair may offer the opportunity to reduce patient risk with less invasive approaches, improve quality of life, and serve to reduce the cost burden. The primary technical safety endpoint is freedom from major adverse events (MAE) at 30 days or during hospitalization if this exceeds 30 days. The primary effectiveness endpoint is the proportion of study subjects with treatment success at 1 year.

ELIGIBILITY:
Inclusion Criteria:

Modified Inclusion Criteria

A patient may be entered into the study if the patient has at least one of the following:

* An aneurysm with a maximum diameter of > 5.5 cm or 2 times the normal diameter just proximal to the aneurysm using orthogonal (i.e., perpendicular to the centerline) measurements
* Aneurysm with a history of growth > 0.5 cm in 6 months
* Saccular aneurysm deemed at significant risk for rupture
* Symptomatic aneurysm greater than 4.5 cm

Other inclusion criteria:

* Axillary or brachial and iliac or femoral access vessel morphology that is compatible with vascular access techniques, devices or accessories, with or without use of a surgical conduit
* Proximal landing zone for the thoracic bifurcation stent graft that has:

  * ≥ 2.5 cm of healthy/nondiseased tissue (including previously placed graft material) (neck) distal to the left subclavian artery (LSA) diameter in the range of 26-42 mm
  * ≥2.5cm of surgical graft distal to the left subclavian artery (LSA) diameter in the range of 26-42mm.
  * Adequate distance from the celiac artery, in order to accommodate cannulation from the antegrade access point when considering the total deployed length of the thoracic bifurcation and visceral manifold
* Minimum branch vessel diameter greater than 5 mm
* Iliac artery distal fixation site, including both native tissue and previously placed graft, greater than or equal to 15 mm in length and diameter in the range of 8 - 25 mm
* Patency of the four major visceral vessels (SMA, celiac, right renal, left renal)
* Age: ≥ 18 years old
* Life expectancy: > 1 year

Exclusion Criteria

General exclusion

* Patient is a good candidate for and elects open surgical repair
* Can be treated in accordance with the instructions for use with a legally marketed endovascular prosthesis
* Is eligible for enrollment in a manufacturer-sponsored investigational device exemption (IDE) at the investigational site
* Unwilling to comply with the follow-up schedule
* Inability or refusal to give informed consent by patient or legal representative
* Patient is pregnant or breastfeeding
* Patient has a contained rupture
* Patient has a ruptured aneurysm
* Patient has a dissection in the treated portion of the aorta
* Obstructive stenting of any or all of the visceral vessels

Medical exclusion criteria

* Known sensitivities or allergies to the materials of construction of the devices, including nitinol (Nickel: Titanium), polyester, platinum-iridium, polytetrafluoroethylene (PTFE), platinum, gold, polyethylene, or stainless steel.
* Known hypersensitivity or contraindication to anticoagulation or contrast media that cannot be adequately medically managed
* Uncorrectable coagulopathy
* Body habitus that would inhibit x-ray visualization of the aorta or exceeds the safe capacity of the equipment
* Patient has had a major surgical or interventional procedure unrelated to the treatment of the aneurysm planned < 30 days of the endovascular repair
* Unstable angina (defined as angina with a progressive increase in symptoms, new onset at rest or nocturnal angina)
* Systemic or local infection that may increase the risk of endovascular graft infection
* Baseline creatinine greater than 2.0 mg/dL
* History of connective tissue disorders (e.g., Marfan Syndrome, Ehler's Danlos Syndrome)

Anatomical exclusion criteria

* Thrombus or excessive calcification within the neck of the aneurysm
* Branch stenosis ≥ 70%
* Anatomy that would not allow maintenance of at least one patent hypogastric artery
* Anatomy that would not allow primary or assisted patency of the left subclavian artery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James H Black, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson J, Nykamp M, Danielson L, Remund T, Kelly PW. A novel endovascular debranching technique using physician-assembled endografts for repair of thoracoabdominal aneurysms. J Vasc Surg. 2014 Nov;60(5):1177-1184. doi: 10.1016/j.jvs.2014.05.090. Epub 2014 Jul 3. PMID 24997805

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Primary Study Arm | Expanded Selection Arm
Started | 2 | 0
Completed | 0 | 0
Not Completed | 2 | 0
Not completed — Death | 2 | 0

BASELINE CHARACTERISTICS:
Population: Enrolled patients who underwent staged/non-staged procedures were analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Primary Study Arm | Expanded Selection Arm | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 0 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Major Adverse Events (MAEs) at 30 Days
Description: Major adverse events include death, bowel ischemia, myocardial infarction, paraplegia, renal failure, respiratory failure, and stroke.
Time Frame: 30 days
Population: Enrolled patients with non-staged, completed procedures were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Study Arm | Expanded Selection Arm
Number analyzed (Participants) | 2 | 0
Participants | 1 | 0

2. Secondary Outcome: Treatment Success at 1 Year
Description: Treatment success is defined as a composite of technical success and freedom from the following:
  Aneurysm enlargement, Aneurysm rupture, Aneurysm-related mortality, Conversion to open repair, Secondary intervention for migration, Type I and III endoleaks, device integrity failure, and patency-related events.
Time Frame: 1 year
Population: Enrolled patients with non-staged, completed procedures were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Study Arm | Expanded Selection Arm
Number analyzed (Participants) | 2 | 0
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: Enrolled patients who received the study intervention were monitored and evaluated for Major Adverse Events (MAEs) and Serious Adverse Events (SAEs).
Arm/Group | Primary Study Arm | Expanded Selection Arm
All-Cause Mortality (participants affected / at risk) | 2/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/0
Other Adverse Events (participants affected / at risk) | 0/2 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Study Arm (N=2) | Expanded Selection Arm (N=0)
bowel ischemia (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Enrollment is permanently closed because the investigational device is no longer manufactured. The target enrollment was not reached and there was insufficient power to measure the effect of the intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT03637374/Prot_SAP_000.pdf